CLINICAL TRIAL: NCT05022953
Title: The Effect of Digital Storytelling on Nursing Students' Compliance With Isolation Precautions and Their Knowledge Levels: A Randomized Controlled Trial
Brief Title: The Effect of Digital Storytelling on Nursing Students' Compliance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Sule BIYIK BAYRAM, Assistant Professor, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KaradenizTU-1
Record Dates: First submitted 2021-08-17; First posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Education; Isolation; Nursing Students
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Story Group (Experimental): Digital Story Group: One of the researchers gave the experimental group participants a 15-minute briefing on how to perform digital storytelling. She also told them not to talk to the control group participants about the content of the briefing. She created a Pixton account (https://edu.pixton.com/educators/) and a class named "Isolation." She sent the link (https://join.pixton.com/x5xb6) to the experimental group participants. She asked them to click on the link and make stories out of their knowledge of isolation in four weeks.
  Interventions: Other: Education, dijital storytelling
- Control Group (No Intervention): Control group participants did not go through any training in isolation.

INTERVENTIONS:
Other: Education, dijital storytelling — Digital story
  Arms: Digital Story Group

SUMMARY:
This study investigated the effect of digital storytelling on nursing students' compliance with isolation precautions and their knowledge levels.This was a pretest-posttest open-label randomized controlled trial. The nursing department of the faculty of health sciences of a university in the eastern Black Sea region of Turkey. The sample consisted of 109 fourth-year nursing students divided into groups of experimental (n=66) and control (n=43). Data were collected using a demographic characteristics questionnaire, an Isolation Knowledge Test (IKT), a Questionnaire of Students' Opinions on Digital storytelling (QSODS), and the Scale of Compliance with Isolation Precautions (SKIP). The experimental group attended a digital storytelling activity (intervention), while the control group received an education based on the curriculum. The data were analyzed using the Mann-Whitney U test, the Wilcoxon test, the Analysis of variance (ANOVA), and the Spearman correlation test.

ELIGIBILITY:
Inclusion Criteria:

* Being voluntary
* Having access to the Internet

Exclusion Criteria:

* Not attending the digital storytelling activity (intervention)
* Not taking the posttest

Ages: 21 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Distribution of students according to descriptive characteristics. | 1 month
  The 11-item demographic characteristics questionnaire was based on a literature review conducted by the researchers (Özden and Özveren, 2016; Orabi, 2017; Sarier and Kurşun, 2020).
  The experimental and control group participants had a mean age of 22.57±2.28 and 21.79±0.80, respectively. The experimental group consisted of 56 women and ten men. The control group consisted of 38 women and six men

SECONDARY OUTCOMES:
The difference between the pre, post and follow-up knowledge scores of the control and experimental group students | 1 month
  The Isolation Knowledge Test (IKT) was based on a literature review conducted by the researchers (Erden et al., 2015, Doğanay et al., 2013, Karabay et al., 2018). Three experts in nursing fundamentals were consulted to develop the test. The draft test consisted of 40 statements. A pilot study was conducted to check for the intelligibility and relevance of the statements and to calculate item difficulty and item discrimination indices.
  was a significant difference between pretest and posttest IKT scores in the experimental group (p=0.01). There was also a significant difference between posttest and follow-up IKT scores in the experimental group (p=0.01). The experimental group had significantly higher follow-up IKT scores than pretest scores.
The difference between the control and experimental group scores according to the total and sub-dimensions of the scale | 2 months
  The Scale of Compliance with Isolation Precautions (SCIP) was developed by Tayran and Ulupınar (2011). The scale consists of 18 items scored on a five-point Likert-type scale ("1 = Strongly disagree," "2 = Disagree," "3 = Neither agree nor disagree," "4 = Agree," "5 = Strongly agree"). The scale has a Cronbach's Alpha of 0.85 (Tayran & Ulupınar, 2011), which was 0.86 (pretest) and 0.78 (posttest) in the present study.
  There was no significant difference in pretest SCIP scores between the experimental and control groups. However, there was a significant difference in posttest SCIP scores between them. The experimental group had significantly higher posttest SCIP scores than pretest scores (p=0.00). It had significantly higher follow-up SCIP scores than posttest and pretest scores. There was no significant difference between the control group's pretest, posttest, and follow-up SCIP scores
The following are quotations from the experimental group participants about digital storytelling. | 2 months
  The Questionnaire of Students' Opinions on Digital Storytelling (QSODS) consisted of three open-ended questions on (1) the contribution of digital storytelling to learning, (2) the effect of digital storytelling on students' compliance with isolation precautions and knowledge levels, and (3) students' opinions about digital storytelling.
  The following are quotations from the experimental group participants about digital storytelling.
  "I realized that I had some gaps in my knowledge of isolation methods and protective measures. It [digital storytelling] helped me fill those gaps." [Student (S). 10].
  I think that it's [digital storytelling] fun and instructive. I helped me go over what I already knew and learn new stuff (S.12).
  We've had distance learning for a long time, so this storytelling thing helped me feel like I was in it" (S. 54).

CONTACTS AND LOCATIONS:
Overall Officials: Emel Gulnar, PhD, Study Chair — Kırıkkale University; Nurcan Caliskan, PhD, Study Chair — Gazi University; Cigdem Torun Kılıc, Msc, Study Chair — Karadeniz Teknik University
Locations (1):
- Sule BIYIK BAYRAM, Trabzon, Turkey (Türkiye)